CLINICAL TRIAL: NCT04071925
Title: 9000 URETHRA STUDY: a Prospective, Observational Study About Urethroplasty for Urethral Stricture Disease
Brief Title: 9000 URETHRA STUDY: a Study About Urethroplasty for Urethral Stricture Disease
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201940616
Record Dates: First submitted 2019-08-12; First posted 2019-08-28 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Urethral Stricture
Keywords: urethral stricture disease; urethral stricture; urethra; urethroplasty
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Urethroplasty — Open reconstructive surgery to restore urethral patency in case of urethral stricture disease.

SUMMARY:
It has been demonstrated that urethroplasty should be considered the gold standard treatment for urethral stricture disease as it yields higher long-term success rates than endoscopic treatment options such as direct vision internal urethrotomy (DVIU) or dilation. Many data about these procedures exist, although most of the publications about urethroplasty are retrospective and involve a tremendous risk of bias. To address these issues, this study is designed to prospectively gain evidence about this matter in all patient subgroups facing a potential treatment with urethroplasty: native men, native women, transmen, transwomen and children.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed written informed consent according to the rules of Good Clinical Practice (Declaration of Helsinki) and national regulations.
* Patient age ≥ 6 years.
* If a patient reaches the age of 18 years, he or she will have to provide a new voluntarily signed written informed consent. All patients reaching the age of 18 years will be contacted by the Principal Investigator or Subinvestigator to provide a new voluntarily signed written informed consent.

Exclusion Criteria:

- Absence of signed written informed consent and thus a patient unwilling to participate.

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Native male and female + transman and transwomen + boys and girls < 18 years old
Study Population: Native men, native women, transmen, transwomen and children with urethral stricture disease.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | From date of surgery until the date of stricture recurrence or date of death from any cause, whichever came first, assessed up to 120 months postoperatively
  Interval between operation and latest follow-up moment at which the patiënt remains failure-free

SECONDARY OUTCOMES:
Change in erectile function | From the date of preoperative questionnaire completion until 24 months postoperatively.
  Assessment preoperatively and postoperatively using the IIEF-5 (International Index of Erectile Function) questionnaire (a 5-item questionnaire, total score on 25, higher score indicating better erectile function).
Change in ejaculatory function | From the date of preoperative questionnaire completion until 24 months postoperatively.
  Assessment preoperatively and postoperatively using the MSHQ-EjD (Male Sexual Health Questionnaire - Ejaculatory Dysfunction) short form questionnaire (a 3-item questionnaire, total score on 15, higher score indicating better ejaculatory function)
Change in urinary function | From the date of preoperative questionnaire completion until 24 months postoperatively.
  Assessment preoperatively and postoperatively using the ICIQ-MLUTS (International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms) module questionnaire (a 6-item questionnaire, total score on 24, higher score indicating more urinary bother)
Change in urinary continence | From the date of preoperative questionnaire completion until 24 months postoperatively.
  Assessment preoperatively and postoperatively using the ICIQ-UI (International Consultation on Incontinence Questionnaire - Urinary Incontinence) short form questionnaire (a 3-item questionnaire, total score on 21, higher score indicating more incontinence).
Change in quality of life | From the date of preoperative questionnaire completion until 24 months postoperatively.
  Assessment preoperatively and postoperatively using the EQ-5D-3L questionnaire (a 5-item questionnaire generating a digit score, each of the 5 items can be scored with 1, 2 or 3 (e.g. 11213), higher digit score indicating lower quality of life).
Change in general quality of life | From the date of preoperative questionnaire completion until 24 months postoperatively.
  Assessment preoperatively and postoperatively using the EQ-VAS (Visual Analogue Scale) (a numeric scale ranging from 0 to 100, higher score indicating better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Lumen, Principal Investigator — University Hospital, Ghent; Marjan Waterloos, Study Chair — University Hospital, Ghent; Wesley Verla, Study Director — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Dept. of Urology, Ghent University Hospital, Ghent
  - University Hospital Ghent, Ghent

IPD SHARING:
Plan to Share IPD: No